CLINICAL TRIAL: NCT03256071
Title: Low Dose Decitabine + Modified BUCY Conditioning Regimen for High Risk Acute Myeloid Leukemia Undergoing Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Jiangsu University (Other); Xuzhou Medical University (Other); Southeast University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAC+BUCY
Record Dates: First submitted 2017-05-21; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloid Leukemia; Allogeneic Hematopoietic Stem Cell Transplantation; Conditioning
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decitabine plus Modified BUCY (Experimental): For high-risk patients with Acute Myeloid Leukemia (AML) undergoing allo-HSCT, The Decitabine plus Modified BuCy regimen consisted of decitabine,semustine,cytarabine, busulfan and cyclophosphamide.
  Interventions: Drug: Decitabine plus Modified BUCY
- Modified BUCY (Active Comparator): For high-risk patients with Acute Myeloid Leukemia (AML) undergoing allo-HSCT, The Modified BuCy regimen consisted of semustine,cytarabine, busulfan and cyclophosphamide.
  Interventions: Drug: Modified BUCY

INTERVENTIONS:
Drug: Decitabine plus Modified BUCY — Decitabine:20 mg/m²/day on day -14 to -10;
  Modified BUCY:
  1. Sibling:semustine 250 mg/m²/day on day -9;cytarabine 2 g/m²/day on day -8；busulfan 3.2mg/kg/day on day -7 to -5;cyclophosphamide 1.8g/m²/day on day -4 to -3.
  2. Unrelated:semustine 250 mg/m²/day on day -10;cytarabine 2 g/m²/day on day -9 to -8；busulfan 3.2mg/kg/day on day -7 to -5;cyclophosphamide 1.8g/m²/day on day -4 to -3.
  3. Haploidentical:semustine 250 mg/m²/day on day -10;cytarabine 4 g/m²/day on day -9 to -8；busulfan 3.2mg/kg/day on day -7 to -5;cyclophosphamide 1.8g/m²/day on day -4 to -3.
  Arms: Decitabine plus Modified BUCY
Drug: Modified BUCY — 1. Sibling:semustine 250 mg/m²/day on day -9;cytarabine 2 g/m²/day on day -8；busulfan 3.2mg/kg/day on day -7 to -5;cyclophosphamide 1.8g/m²/day on day -4 to -3.
  2. Unrelated:semustine 250 mg/m²/day on day -10;cytarabine 2 g/m²/day on day -9 to -8；busulfan 3.2mg/kg/day on day -7 to -5;cyclophosphamide 1.8g/m²/day on day -4 to -3.
  3. Haploidentical:semustine 250 mg/m²/day on day -10;cytarabine 4 g/m²/day on day -9 to -8；busulfan 3.2mg/kg/day on day -7 to -5;cyclophosphamide 1.8g/m²/day on day -4 to -3.
  Arms: Modified BUCY

SUMMARY:
The purpose of this prospective, open-label, randomized multicenter study is to evaluate the safety and efficacy of low dose decitabine in combination with modified BUCY vs modified BUCY as a myeloablative conditioning regimen for high-risk patients with acute myeloid leukemia (AML) undergoing allogeneic hematopoietic stem cell transplantation (Allo-HSCT).

DETAILED DESCRIPTION:
Allo-HSCT is the most effective treatment stratagey for high risk acute myeloid leukemia. At present, modified BUCY is the standard conditioning regimen for AML undergoing allo-HSCT in our institute. However, relapse occured in as high as 30-50% high risk AML patients after allo-HSCT. Thus, the best conditioning regimen for this subgroup remains to be optimized. Low dose decitabine in combination with chemotherapy have been shown to improve comple remission rate of high risk AML patients. To reduce the relapse rate after allo-HSCT, low dose decitabine is added in the modified BUCY regimen. In this study, the safety and efficacy of low dose decitabine + modified BUCY vs modified BUCY myeloablative conditioning regimens in high risk undergoing allo-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 60 years.
* Diagnosis of high-risk acute myeloid leukemia at the time of transplant. ("High-risk" AML features are defined by the following: relapsed or primary refractory AML; Secondary AML（AML Secondary to myelodysplastic syndrome(MDS) or treatment-related AML); extramedullary leukemia; adverse cytogenetic abnormalities of monosomy 5, monosomy 7, or deletion of 5q; or presence of FLT3 positive internal tandem duplication (FLT3/ITD+), particularly high allelic ratio.)
* Patient must have adequate pre-transplant organ function.

Exclusion Criteria:

* Age <12 or >60 years.
* Uncontrolled bacterial, viral, fungal, or other infection before conditioning regimen.
* Any other severe concurrent diseases, or have a history of serious organ dysfunction.
* Pregnant or lactating females.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 year
  time from randomization to the first of reccurrence or death
overall survival (OS) | 3 year
  time from randomization to death from any cause

SECONDARY OUTCOMES:
veno-occlusive disease (VOD) | 3 year
  incidence of veno-occlusive disease (VOD) events
graft-versus-host disease (GvHD) | 3 year
  incidence and severity of acute (aGvHD) and chronic graft-versus-host disease (cGvHD)
transplant related mortality （TRM） | 3 year
  cumulative incidence of transplant related mortality
relapse | 3 year
  cumulative incidence of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China